CLINICAL TRIAL: NCT00627627
Title: A Phase 2, Open-Label, Single-Arm, Multicenter, Multinational Study to Evaluate the Antitumor Activity and Safety of IPI-504, A Novel Small Molecule Inhibitor of Heat Shock Protein 90(HSP90), in Patients With Locally Advanced or Metastatic Human Epidermal Growth Factor Receptor 2-Positive(HER2+) Breast Cancer That Has Progressed Despite Prior Her2=Targeted Therapy
Brief Title: A Study to Evaluate the Antitumor Activity and Safety of IPI-504 in Patients With Advanced Breast Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Redirect focus of the indication
Sponsor: MedImmune LLC (Industry)
Responsible Party: David E. Weng, M.D., Ph. D., MedImmune Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP153
Record Dates: First submitted 2008-02-21; First posted 2008-03-03 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — tanespimycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): IPI-504
  Interventions: Drug: IPI-504

INTERVENTIONS:
Drug: IPI-504 — dose of 400 mg/m2 as a 30-60 minute IV infusion as part of a 21-day treatment cycle

SUMMARY:
To evaluate the antitumor activity following treatment with IPI-504 in patients with breast cancer.

DETAILED DESCRIPTION:
To evaluate the antitumor activity following treatment with IPI-504 in patients with locally advanced or metastatic HER2+ breast cancer that has progressed despite prior HER2-targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult women at least 18 years of age at the time of signing the Informed Consent Form;
* Written informed consent and HIPAA authorization (applies to covered entities in the USA only) obtained from the patient prior to performing any study-related procedures, including screening visits;
* Pathologically confirmed breast cancer from assessment of primary or metastatic breast cancer;
* Locally advanced or metastatic breast cancer as defined as a T4 primary tumor and Stage IIIB/ IIIC disease or Stage IV disease, respectively, according to the Sixth Edition of the American Joint Committee on Cancer [AJCC] TNM System (Appendix A);
* Measurable disease according to RECIST - lesions that can be accurately measured in at least one dimension with longest diameter ³ 20 mm using conventional computed tomography (CT) or magnetic resonance imaging (MRI) scan or ³ 10 mm with spiral CT scan; the use of chest x-ray is not encouraged, however, it may be used if necessary;
* HER2-expressing primary or metastatic tumor (Grade 3+ staining intensity [on a scale of 0 to 3] via IHC assays or HER2 amplification on fluorescence in situ hybridization), with results of the most recent biopsy taken as indicative of HER2 status;
* Progression after treatment with at least 1 but not more than 3 regimens containing trastuzumab or lapatinib (treatment regimens that do not include trastuzumab or lapatinib do not qualify) for adjuvant, neoadjuvant, locally advanced, or metastatic disease with either one of the following stipulations:

  1. Patients may have received neoadjuvant or adjuvant treatment with prior trastuzumab or lapatinib treatment but must have demonstrated no evidence of disease progression for >12 months following completion of therapy;
  2. Patients have received a trastuzumab-based therapy for locally advanced or metastatic disease for a minimum of 9 weeks duration. Patients may have received more than 1 trastuzumab-based combination therapy; Patients have received a lapatinib-based therapy for locally advanced or metastatic diseases for a minimum of 9 weeks duration;
* Resolution of all toxic side effects of prior chemotherapy, radiotherapy or surgical procedures to NCI CTCAE Grade ≤ 1 or patient's baseline;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 (see Appendix B);
* Life expectancy of at least 3 months;
* Left ventricular ejection fraction > 45%;
* Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3; platelet count ≥ 100,000 cells/mm3; hemoglobin ≥ 9.0 g/dL (may be increased to this level with transfusion as long as there is no evidence of active bleeding);
* Prothrombin time or international normalized ratio within normal range (unless a patient is receiving anticoagulation therapy), or PTT within normal range;
* AST and ALT ≤ 2.5 ´ upper limit of normal (ULN) or ≤ 5 ´ ULN for patients with liver metastases; total bilirubin ≤ 1.5 ´ ULN [unless due to Gilbert's syndrome (unconjugated hyperbilirubinemia) in which case the bilirubin should be < 3.5mg/dL); hepatic alkaline phosphatase ≤ 2.5 ´ ULN;
* Serum creatinine ≤ 1.5 ´ ULN and calculated creatinine clearance ≥ 30 mL/min;
* Women with central nervous system (CNS) metastases are eligible if they are clinically stable for at least 3 months after the discontinuation of prior corticosteroid therapy;
* Female patients must be of non child-bearing potential or using effective contraception, eg, use of oral contraceptives with an additional barrier method (since the study drug may impair the effectiveness of oral contraceptives), double barrier methods (diaphragm with spermicidal gel or condoms with contraceptive foam), Depo-Provera, partner vasectomy, total abstinence, and willing to continue the effective contraception method for 30 days after the last dose of IPI-504; and
* Patients must be able to adhere to the study visit schedule and all protocol requirements.

Exclusion Criteria:

* Previous treatment with 17-AAG, 17-DMAG, or other known Hsp90 inhibitor;
* Concurrent radiation or surgery therapy;
* Treatment for breast cancer with any approved or investigational product, including any local or systemic therapy within 4 weeks prior to first dose of IPI-504 in this study;
* Initiation or discontinuation of concurrent medication that alters CYP3A activity within 2 weeks prior to treatment with IPI-504. Patients who are on a stable dose of drugs known to alter CYP3A activity for > 2 weeks are eligible to enroll;
* Presence of active infection or systemic use of antimicrobials within 72 hours prior to treatment with IPI-504;
* Untreated brain metastases (patients with a history of brain metastases are eligible as long as definitive treatment has been given and patients are clinically stable for at least 3 months after the discontinuation of prior corticosteroid therapy);
* Significant co-morbid condition or disease which in the judgment of the Investigator would place the patient at undue risk or interfere with the study (eg, cardiac disease such as acute coronary syndrome or unstable angina within 6 months, uncontrolled hypertension, arrhythmia requiring medication or mechanical control, conduction system abnormality such as left bundle branch block or second degree heart block, cirrhotic liver disease, cerebrovascular accident, or other conditions);
* Women who are pregnant or lactating;
* Sinus bradycardia (resting heart rate < 50 bpm) secondary to intrinsic conduction system disease; Patients with sinus bradycardia secondary to pharmacologic treatment may enroll if withdrawal of the treatment results in normalization of the resting heart rate to within normal limits;
* Screening QTc > 470 msec, or previous history of QTc prolongation while taking other medications; or
* Active or recent history (within 3 months) of keratitis or keratoconjunctivitis.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the antitumor activity, assessed by ORR which will be determined using RECIST, following treatment with IPI-504 in patients with locally advanced or metastatic HER2+ breast cancer that has progressed despite prior HER2-targeted therapy. | 30 days after discontinuation of IPI-504

SECONDARY OUTCOMES:
To evaluate other antitumor activities, safety, and PK parameters of IPI-504 in this patient population. | 30 days after discontinuation of IPI-504

CONTACTS AND LOCATIONS:
Overall Officials: David E. Weng, M.D., PhD, Study Director — MedImmune LLC
Locations (7):
- United States (7):
  - Georgetown Univ Medical Cntr, Lombardi Comprehensive Cancer Center,, Washington D.C., District of Columbia
  - Lynn Regional Cancer - West Campus, Boca Raton, Florida
  - Medical Specialists of the Palm Beaches, Lake Worth, Florida
  - "Duke University Med Cntr Breast Oncology Research Program, Durham, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic Medical Center, Cleveland, Ohio
  - Low County Hen/Onc, Mt. Pleasant, South Carolina